CLINICAL TRIAL: NCT05760612
Title: A Randomized, Open-Label, Phase III Trial Comparing Adjuvant Trastuzumab Plus Neratinib Versus Trastuzumab Plus Pertuzumab in Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer With Residual Cancer Burden 0/I After Neoadjuvant Trastuzumab Plus Pertuzumab
Brief Title: Adjuvant Trastuzumab Plus Neratinib in Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer After Neoadjuvant Trastuzumab Plus Pertuzumab
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, Chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-075-03
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Early-stage Breast Cancer; HER2-positive Breast Cancer; Adjuvant Treatment After Trastuzumab; RCB Classification 1-2; Neratini
Keywords: Hormone receptor positive HER2 positive breast cancer; targeted therapy; adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; neratinib; pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab combined with Pertuzumab (Active Comparator): Trastuzumab (8 mg/kg IV loading dose, followed by 6 mg/kg IV once every 3 weeks), and pertuzumab (840 mg IV loading dose, followed by 420 mg IV once every 3 weeks). This regimen will be repeated for a total of 18 cycles,encompassing both the preoperative and adjuvant phases.
  Interventions: Drug: Trastuzumab and Pertuzumab
- Trastuzumab combined with neratinib (Experimental): Trastuzumab (8 mg/kg IV loading dose, followed by 6 mg/kg IV once every 3 weeks), and neratinib 240 mg orally once daily. The trastuzumab treatment will be continued for a total of 18 cycles, encompassing both the preoperative and adjuvant phases, while neratinib will be maintained throughout the adjuvant period.
  Interventions: Drug: Trastuzumab and neratinib

INTERVENTIONS:
Drug: Trastuzumab and neratinib — Trastuzumab (8 mg/kg IV loading dose, followed by 6 mg/kg IV once every 3 weeks), and neratinib 240 mg orally once daily. The trastuzumab treatment will be continued for a total of 18 cycles, encompassing both the preoperative and adjuvant phases, while neratinib will be maintained throughout the adjuvant period.
  Arms: Trastuzumab combined with neratinib
Drug: Trastuzumab and Pertuzumab — Trastuzumab (8 mg/kg IV loading dose, followed by 6 mg/kg IV once every 3 weeks), and pertuzumab (840 mg IV loading dose, followed by 420 mg IV once every 3 weeks). This regimen will be repeated for a total of 18 cycles,encompassing both the preoperative and adjuvant phases.
  Arms: Trastuzumab combined with Pertuzumab

SUMMARY:
Neratinib is an irreversible pan-HER tyrosine kinase inhibitor (TKI). Currently, no studies have investigated the use of macromolecular anti-HER2 agents combined with TKIs for the treatment of non-pCR HER2-positive breast cancer following neoadjuvant therapy. Furthermore, there are no prospective randomized controlled trials comparing trastuzumab plus pertuzumab versus trastuzumab plus TKIs in HER2-positive breast cancer patients with residual cancer burden class (RCB) I or II after neoadjuvant trastuzumab and pertuzumab. Therefore, this study aimed to evaluate the efficacy and safety of adjuvant trastuzumab plus neratinib in patients with hormone receptor-positive/HER2-positive breast cancer and RCB 0/I following neoadjuvant trastuzumab and pertuzumab therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years;
2. Eastern Cooperative Oncology Group performance status of 0 or 1;
3. Clinical stage at initial diagnosis (per the 8th edition of the American Joint Committee on Cancer Staging Manual): cT1-4/N1-3/M0 (cT1mi/N0 or cT1a-b/N0 are eligible), meeting the criteria for neoadjuvant therapy as per NCCN 2022 guidelines;
4. Histologically confirmed hormone receptor-positive (estrogen receptor ≥1% and/or progesterone receptor ≥1%) and HER2-positive (immunohistochemistry 3+ or fluorescence in situ hybridization-positive) invasive breast cancer;
5. Completion of ≥4 cycles of neoadjuvant therapy with trastuzumab and pertuzumab, without recurrence or metastatic disease prior to adjuvant treatment; residual cancer burden class 0 or I after neoadjuvant therapy; time from initial surgery to randomization ≤12 weeks;
6. Adequate organ function within 2 weeks prior to screening (without transfusion or use of growth factors):

   * Absolute neutrophil count ≥1.5 × 10⁹/L;
   * Platelet count ≥90 × 10⁹/L;
   * Hemoglobin ≥90 g/L;
   * Total bilirubin ≤1.5 × upper limit of normal (ULN);
   * Alanine aminotransferase and aspartate aminotransferase ≤1.5 × ULN;
7. Post-neoadjuvant therapy echocardiography showing left ventricular ejection fraction (LVEF) ≥50% during screening, with an absolute decrease of ≤15% compared to pre-chemotherapy values; if no pre-chemotherapy LVEF assessment is available, LVEF must be ≥55% during screening;
8. Life expectancy ≥6 months;
9. For premenopausal or non-sterilized female patients: agreement to abstain from sexual activity or use effective non-hormonal contraception during study treatment and for 8 weeks after the last dose;
10. Willingness to participate voluntarily, provide signed informed consent, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. History of local or regional breast cancer recurrence;
2. Clinical stage IV (metastatic) breast cancer;
3. Bilateral breast cancer;
4. History of other malignant tumors within the past 5 years, except for curatively treated cervical carcinoma in situ, basal cell carcinoma, or cutaneous squamous cell carcinoma;
5. Prior treatment with pyrotinib, lapatinib, neratinib, or other tyrosine kinase inhibitors; trastuzumab emtansine; or any antitumor biological or immunotherapy;
6. Concurrent participation in another clinical trial involving antitumor therapy, including endocrine therapy, bisphosphonate therapy, or immunotherapy;
7. Significant cardiac disease, including:

   * Heart failure or systolic dysfunction (LVEF < 50%);
   * Poorly controlled arrhythmias (e.g., atrial tachycardia, significant ventricular arrhythmia, or high-grade atrioventricular block);
   * Angina requiring antianginal medication;
   * Clinically significant valvular heart disease;
   * Electrocardiographic evidence of transmural myocardial infarction;
   * Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg) despite medication;
8. Impaired drug absorption due to dysphagia, intestinal obstruction, or other gastrointestinal disorders;
9. History of neurological or psychiatric conditions that may compromise compliance or informed consent;
10. Chronic gastrointestinal disorders with predominant diarrhea;
11. Known hypersensitivity to any study drug components; history of immunodeficiency (e.g., HIV positivity, congenital or acquired immunodeficiency disorder), or prior organ transplantation;
12. Pregnancy, lactation, or positive pregnancy test at baseline in women of childbearing potential;
13. Severe comorbidities that may interfere with treatment, including active infections (e.g., hepatitis B, hepatitis C, tuberculosis, syphilis) or any other condition deemed by the investigator to render the patient unsuitable for trial participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2028-02-16 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Invasive disease free survival, IDFS | During the 3 years after random assignment
  The time from random assignment until the first occurrence of invasive disease recurrence, distant recurrence, or death from any cause.

SECONDARY OUTCOMES:
Disease free survival, DFS | During the 3 years after random assignment
  The time from random assignment until recurrence, the development of a second cancer, or death from any cause.
Overall survival, OS | During the 3 years after random assignment
  The time from randomization to death from any cause.
Distant disease free survival, DDFS | During the 3 years after random assignment
  The time from random assignment until the first occurrence of distant recurrence or death from any cause.
Incidence and severity of adverse events | From signing the informed consent form until 28 days after completion of adjuvant treatment
  The incidence and severity of adverse events will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Sun Yat-sen Memorial Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No